CLINICAL TRIAL: NCT04560478
Title: THE EFFICACY OF MI VARNISH VERSUS PRO SEAL SEALANT ON PREVENTION OF WHITE SPOT LESIONS IN ORTHODONTIC PATIENTS: A RANDOMIZED CLINICAL TRIAL
Brief Title: Comparing Fluoride Varnish and Sealant to Prevent White Spots in Orthodontic Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Texas A&M University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: COD_Ortho2
Record Dates: First submitted 2020-09-17; First posted 2020-09-23 (Actual); Last update posted 2020-09-23 (Actual); Status verified 2020-09

CONDITIONS: White Spot Lesion
Keywords: Oral Hygiene; Orthodontics; White spot lesion; enamel decalcification

STUDY DESIGN:
Intervention Model Description: single center, parallel, randomized clinical trial
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Pro Seal Sealant (Active Comparator): ProSeal Sealant was applied to the facial surfaces of the maxillary anterior teeth (canine to canine)
  Interventions: Device: Pro Seal Sealant
- MI Varnish (Active Comparator): MI Fluoride Varnish was applied to the maxillary anterior teeth (canine to canine)
  Interventions: Device: MI Varnish

INTERVENTIONS:
Device: Pro Seal Sealant — Sealant was reapplied every 3 months
  Arms: Pro Seal Sealant
Device: MI Varnish — Fluoride varnish was applied every 4-6 weeks
  Arms: MI Varnish

SUMMARY:
The purpose of the study is o compare the efficacy of CPP-ACP MI Varnish and ProSeal sealant in preventing white spot lesion (WSL) formation in orthodontic patients.

DETAILED DESCRIPTION:
This prospective randomized clinical trial included 40 orthodontic patients between the ages of 12-17 who were randomly allocated to two groups. Group 1 (Sealant Group) received sealant on the maxillary anterior canines, lateral incisors, and central incisors, with reapplication of the sealant every 3 months. Group 2 (Varnish Group) had MI Varnish applied every 4-6 weeks, without sealant placed on the maxillary anterior teeth. White spot lesion formation was evaluated with standardized digital photographs at two timepoints, T1 (initial appointment before bonding), and T2 (12 months later, with brackets removed). The brackets were removed in order to facilitate an adequate photographic exam. Photographs were analyzed side-by-side at the conclusion of the study with the Enamel Decalcification Index (EDI). The location of WSLs were recorded by tooth type and by region. Oral hygiene was evaluated at T1 and T2.

ELIGIBILITY:
Inclusion Criteria:

* no significant medical history
* no underlying medical problems such as Sjogren's Syndrome or conditions requiring more than 2 medications (to prevent bias of possible dry mouth)
* less than 17 years old at the start of orthodontic treatment,
* fully erupted permanent maxillary canines and incisors, starting fixed orthodontic treatment
* ability to come to appointments every 4-6 weeks.

Exclusion Criteria:

* professional fluoride application in the last 3 months
* allergy to milk
* untreated cavitated lesions
* heavy initial fluorosis
* dry mouth
* pregnancy
* any illness/condition that the investigators felt would affect the study outcome.

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 40 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2020-02-10 (Actual); Study Completion 2020-03-01 (Actual)

PRIMARY OUTCOMES:
Enamel Decalcification Index | 12 months
  Extent and severity of white spot lesion formation

SECONDARY OUTCOMES:
Location of White Spot Lesions | 12 months
  Mesial, Distal, Incisal or Gingival Region
Most Common Tooth for White Spot Formation | 12 Months
  Maxillary Canine, Lateral, or Central Incisor
Oral Hygiene Status | 12 Months
  Measurement of plaque accumulation on maxillary teeth
Sex Differences | 12 Months
  Male versus Female

CONTACTS AND LOCATIONS:
Overall Officials: Peter Buschang, PhD, Principal Investigator — Texas A&M University
Locations (1):
- Texas A&M University College of Dentistry, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No
Individual results of the study will not be shared.

REFERENCES:
- [Result] Banks PA, Richmond S. Enamel sealants: a clinical evaluation of their value during fixed appliance therapy. Eur J Orthod. 1994 Feb;16(1):19-25. doi: 10.1093/ejo/16.1.19. PMID 8181546
- [Result] Turesky S, Gilmore ND, Glickman I. Reduced plaque formation by the chloromethyl analogue of victamine C. J Periodontol. 1970 Jan;41(1):41-3. doi: 10.1902/jop.1970.41.41.41. No abstract available. PMID 5264376